CLINICAL TRIAL: NCT00790465
Title: Efficacy of Dark Chocolate in Achalasia Patients: Placebo-Controlled Study
Brief Title: Efficacy of Dark Chocolate in Achalasia Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Dr. Guy Rosner, gastroenterologist, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: TASMC-08-GR-370-CTIL; achalasia1
Record Dates: First submitted 2008-11-12; First posted 2008-11-13 (Estimated); Last update posted 2008-11-13 (Estimated); Status verified 2008-11

CONDITIONS: Achalasia
Keywords: achalasia; lower esophageal sphincter; nitric oxide; dark chocolate; flavanols
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): dark chocolate consumption during manometry and 2 weeks treatment with dark chocolate
  Interventions: Dietary Supplement: dark chocolate
- 2 (Other): placebo comparator: 7 grams of placebo-chocolate at day 1 during manometry, and than crossover to treatment with dark chocolate for 2 weeks.
  Interventions: Dietary Supplement: placebo chocolate with crossover to dark chocolate

INTERVENTIONS:
Dietary Supplement: dark chocolate — 21 g/d of dark chocolate for 2 weeks (7 g. before each meal). 7 grams of dark chocolate at day 1 during manometry.
  Other Names: FruiBel chocolate, Belgium.
  Arms: 1
Dietary Supplement: placebo chocolate with crossover to dark chocolate — Placebo at day 1 during manometry, and than crossover to dark chocolate for 2 weeks treatment.
  Other Names: FruiBel chocolate, Belgium
  Arms: 2

SUMMARY:
Flavanols, present in dark chocolate, were shown to induce Nitric Oxide synthesis. Since Nitric Oxide facilitates smooth muscle relaxation, it might ease the relaxation of the LES (lower esophageal sphincter)as well.

The objective of the present study is to evaluate tha efficacy of dark chocolate in improving LES relaxation in achalasia patients.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of "achalasia"
* "Achalasia" diagnosis during manometry at day 1 of the study.

Exclusion Criteria:

* pregnancy
* pseudoachalasia
* consumption of GI-motility modifiers durin 72 hours preceding the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-11 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Lower Esophageal Sphincter relaxation before and after dark chocolate consumption. | day 1

SECONDARY OUTCOMES:
achalasia symptoms before and during dark-chocolate consumption | 2 weeks